CLINICAL TRIAL: NCT02409407
Title: Effectiveness of Oral Versus Vaginal Misoprostol Before Office Hyteroscopy in Infertile Patients
Brief Title: Misoprostol Before Hysteroscopy in Infertile Cases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Yomna Ali Bayoumi, Lecturer of Obstetrics and Gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MS20150303
Record Dates: First submitted 2015-04-01; First posted 2015-04-06 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Misoprostol

ARMS (3):
- Oral Misoprostol (Experimental): oral misoprostol ( prostaglandins E1 analogue) will be administered at a dose of 600 µg (200 µg every 8 hours), starting 24 hours before office hysteroscopy.
  Interventions: Drug: Misoprostol , Prostaglandins E1 analogue
- Vaginal Misoprostol (Experimental): vaginal misoprostol ( prostaglandins E1 analogue)will be administered at a dose of 400 µg (200 µg 12 hours apart, starting 24 hours before office hysteroscopy)
  Interventions: Drug: Misoprostol , Prostaglandins E1 analogue
- Placebo (Placebo Comparator): oral placebo (one pill every 8 hours) will be administered starting 24 hours before the office hysteroscopy.

INTERVENTIONS:
Drug: Misoprostol , Prostaglandins E1 analogue
  Other Names: Misotac
  Arms: Oral Misoprostol; Vaginal Misoprostol

SUMMARY:
The role of hysteroscopy in infertility investigation is to detect possible intrauterine changes that could interfere with implantation or growth or both of the conceptus, with the invention of miniature hysteroscope, it is possible to perform hysteroscopy in an office setting (Outpatient hysteroscopy; OH), for diagnostic and certain therapeutic intervention. It is currently acknowledged as the 'gold standard' investigation of the intrauterine abnormalities.

Cervical priming prior to diagnostic hysteroscopy softens the cervix and lessens the force needed for dilation, thereby potentially reducing the probability of procedural complication such as uterine perforation, cervical laceration, failure to dilate, and creation of a false track that can occur during cervical entry.

Misoprostol is a prostaglandin El analogue, that can be administered either orally or vaginally, that can cause cervical ripening by inducing collagenolytic activity and synthesis of proteoglycans.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged from 20 to 40 years old.
* They are complaining with primary or secondary infertility.
* They undergo investigations including husband semen analysis, hormonal assay, U/S, Hystrosalpingography.

Exclusion Criteria:

* Known sensitivity to misoprostol.
* Any systemic disease contraindicating the use of prostaglandins (cardiovascular disease, hypertension, renal failure, etc).
* Concomitant neurologic disease that could affect the correct evaluation of pain.
* Pregnancy.
* Any contraindication to hysteroscopy such as Pelvic inflammatory disease (PID).
* Heavy uterine bleeding.
* Any uterine abnormality such as pinhole cervix that would obviate passage of a catheter through the cervix.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
level of pelvic pain according to a 10-point visual analogue scale (VAS) | 10 months
  The level of pelvic pain will be rated according to a 10-point visual analogue scale (VAS). The VAS will be applied immediately after the procedure ended

CONTACTS AND LOCATIONS:
Overall Officials: Yomna A Bayoumi, MD, Principal Investigator — Kasr El Aini Hospital
Locations (1):
- Kasr el Ainy hospital, Cairo, Cairo Governorate, Egypt